CLINICAL TRIAL: NCT05649826
Title: Optimization of an Ultrasound Cardiac Guidance Tool
Brief Title: Automated Ultrasound Cardiac Guidance Tool
Status: Recruiting | Type: Observational
Sponsor: UltraSight (Industry)
Responsible Party: Sponsor
Other Study IDs: 002-30 US
Record Dates: First submitted 2022-04-03; First posted 2022-12-14 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Ultrasound Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research examines echocardiography images taken from cardiac patients in relation to the guidance tool developed

DETAILED DESCRIPTION:
The study is an open label, single arm prospective study. This goal of the study is to learn about echocardiography images in relation to the developed guidance tool software in cardiac patients population. Participants will undergo one session of transthoracic echocardiography exam. The ultrasound will be performed by a sonographer for images acquiring purposes

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, aged 18 years and older
2. Subject willing and able to give written informed consent

Exclusion Criteria:

1. Emergency (non-elective) admission within 24 h prior to participating in the study
2. Female subjects who are pregnant (women of childbearing potential will provide a statement that they are not pregnant incorporated in the ICF
3. Unable to lie as required in all the classic positions for standard TTE exam: supine on back / left decubitus
4. Subjects who currently participate in a clinical trial, involving interventional cardiac devices.
5. Subjects who have prior Echo exam with description of Low/Poor quality exam in the echo report.
6. Subjects with BMI above 40.
7. Subjects experiencing a known or suspected acute cardiac event.
8. Subjects with severe chest wall deformity as per previous medical records and physical examination.
9. Subjects who have undergone pneumonectomy.
10. Subjects whose anatomy does not lend itself to yield diagnosable standard echocardiography clips (i.e., situs inversus with dextrocardia, single ventricle anatomy due to congenital heart disease, etc.).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 200 subjects will be enrolled in this study, at least 35% females and 35% males.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Acquisition of transthoracic echocardiography media from up to 200 subjects | up to 5 year
  Several echocardiography views will be acquired from the participants, with in several acoustic windows and views

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ehrman, MD, Principal Investigator — Wayne University Emergency medicine; Noa Avisar, PhD, Study Director — UltraSight
Locations (1):
- Wayne University, Detroit, Michigan, United States